CLINICAL TRIAL: NCT01931657
Title: Pre-treatment With Mifepristone in Patients With Mirena for Optimizing Bleeding Pattern in Pre-menopausal Women
Brief Title: Pretreatment With Mifepristone Prior to Mirena Insertion
Acronym: MiMi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W2009M
Record Dates: First submitted 2013-08-25; First posted 2013-08-29 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Women in Need of Long Acting Reversibel Cntraception With the Intrauterine Levonorgestrel Releasing System, Mirena
Keywords: LNG-IUS; Mirena; Contraception; Bleeding; Hormonal effects in the breast
MeSH Terms: conditions — Hemorrhage | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone prior to Mirena (Experimental): Pretreatment with mifepristone prior to Mirena insertion
  Interventions: Drug: Mifepristone prior to Mirena
- Placebo prior to Mirena (Placebo Comparator): Pretreatment with placebo prior to Mirena insertion
  Interventions: Drug: Placebo prior to Mirena insertion

INTERVENTIONS:
Drug: Mifepristone prior to Mirena
  Other Names: Mifepristone
  Arms: Mifepristone prior to Mirena
Drug: Placebo prior to Mirena insertion
  Arms: Placebo prior to Mirena

SUMMARY:
Hypothesis: Pretreatment with mifeprsitone prior to Mirena placement will induce amenorrhea and reduce bleeding irrregularities during the initial months of Mirena use.

DETAILED DESCRIPTION:
The levonorgestrel releasing intrauterine system (IUS), Mirena, represents a highly effective contraceptive method that is cost-effective and requires limited patient effort. Furthermore Mirena offers numerous noncontraceptive benefits and addresses different medical needs for women in reproductive and non reproductive age. Side effects such as menstrual abnormalities are important reasons for early discontinuation of a contraceptive method. Irregular bleeding pattern and spotting represents a well known adverse effect during the first months of use with Mirena and corresponds to the most important factor that negatively influences the acceptability of the IUS. Up to today no standard treatment has been suggested to resolve this issue.

By inducing amenorrhea within a short period of treatment with an anti-progesterone, mifepristone, prior to insertion of Mirena, the bleeding irregularities during the first months of use might be reduced and could therefore represent an important strategy for increasing acceptability of this contraceptive system.

The purpose of the present study is to evaluate the bleeding pattern during the first months of use of Mirena in patients treated with mifepristone compared to placebo in women using Mirena for contraception. The study will also address the effect of mifepristone on endometrial morphology and breast tissue.

ELIGIBILITY:
Inclusion criteria:

* Pre-menopausal women, >/= 18 years of age.
* Desire of Mirena for contraception
* Good general health (as judged by; general physical examination
* Willing and able to participate after giving informed consent

Exclusion criteria:

* Any hormonal treatment or IUD use within 2 months prior to study start
* History of malignant disorder of the breast
* Any contraindication to mifepristone
* Pregnancy or breast feeding within 2 months prior to study start

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Days with bleeding and spotting | During the first 3 months of Mirena use
  To study the effect of pre-treatment with mifepristone on the initial bleeding pattern in women using LNG-IUS (Mirena)

SECONDARY OUTCOMES:
Endometrial changes | 3 months post Mirena insertion
  To study the effect of mifepristone pre treatment on the endometrium in women before and during treatment with Mirena with special regard to progesteron receptor modulator associated endometrial changes observed following continuos treatment with mifeprsitone (PAEC).
Effects on breast tissue | Evaluated at end of mifeprsitone treatment
  Breast biopsies are obtained at baseline and following 2 months treatment with mifepristone

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden